CLINICAL TRIAL: NCT00405756
Title: A Phase III, Multicentre, Randomized, Double-Blind, Placebo-Controlled, 3-Arm Parallel Group Study To Determine The Efficacy And Safety Of Lenalidomde (Revlimid®) In Combination With Melphalan And Prednisone Versus Placebo Plus Melphalan And Prednisone In Subjects With Newly Diagnosed Multiple Myeloma Who Are 65 Years Of Age Or Older
Brief Title: A Study to Compare MPR With MP in Newly Diagnosed Multiple Myeloma Subjects 65 Years Old or Older.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-MM-015; 2006-001865-41 (EudraCT Number)
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Newly Diagnosed Multiple Myeloma
Keywords: Newly Diagnosed Multiple Myeloma; Celgene; CC-5013; Revlimid; Lenalidomide; Melphalan; Prednisone; Elderly
MeSH Terms: interventions — Lenalidomide; Melphalan; Prednisone; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MPR+R (Experimental): Double-blind induction therapy with melphalan/prednisone and lenalidomide 10 mg (MPR) for up to 9 cycles, followed by maintenance therapy with single-agent lenalidomide (R) 10mg from cycle 10 to disease progression. Optional open-label extension therapy with lenalidomide up to 25 mg for participants with progressive disease.
  Interventions: Drug: Lenalidomide: Double-blind Induction; Drug: Melphalan; Drug: Prednisone; Drug: Aspirin; Drug: Lenalidomide: Double-blind Maintenance; Drug: Lenalidomide: Open-label
- MPR+p (Experimental): Double-blind induction therapy with melphalan/prednisone and lenalidomide 10mg (MPR) for up to 9 cycles, followed by maintenance therapy with placebo (p) from cycle 10 to disease progression. Optional open-label extension therapy with lenalidomide up to 25 mg for participants with progressive disease.
  Interventions: Drug: Lenalidomide: Double-blind Induction; Drug: Melphalan; Drug: Prednisone; Drug: Aspirin; Drug: Placebo; Drug: Lenalidomide: Open-label
- MPp+p (Other): Double-blind induction therapy with melphalan/prednisone and placebo (MPp) for up to 9 cycles, followed by maintenance therapy with placebo (p) from cycle 10 to disease progression. Optional open-label extension therapy with lenalidomide up to 25 mg for participants with progressive disease.
  Interventions: Drug: Melphalan; Drug: Prednisone; Drug: Aspirin; Drug: Placebo; Drug: Lenalidomide: Open-label

INTERVENTIONS:
Drug: Lenalidomide: Double-blind Induction — Double-blind Induction: the starting lenalidomide oral dosing regimen was 10 mg once daily on Days 1 through 21 of each 28 day cycle for up to 9 cycles. Dose was reduced if needed due to dose-limiting toxicity.
  Other Names: Revlimid
  Arms: MPR+R; MPR+p
Drug: Melphalan — Double-blind Induction: the starting melphalan oral dosing regimen in all 3 treatment arms was 0.18 mg/kg daily on Days 1 through 4 of each 28-day cycle for up to 9 cycles. Dose was reduced if needed due to dose-limiting toxicity.
  Other Names: Alkeran
Drug: Prednisone — Double-blind induction: the starting prednisone oral dosing regimen in all 3 treatment arms was 2 mg/kg daily on Days 1 through 4 of each 28-day cycle for up to 9 cycles. Dose was reduced if needed due to dose-limiting toxicity.
Drug: Aspirin — Double-blind induction: low-dose aspirin 75 mg to 100 mg daily for all treatment arms.
  Double-blind maintenance: at the investigator's discretion
Drug: Placebo — Double-blind induction: participants in treatment arm MPp+p received placebo once daily on Days 1 through 21 of each 28-day cycle for up to 9 cycles.
  Double-blind maintenance: participants in treatment arms MPR+p and MPp+p received placebo once daily on Days 1 through 21 of each 28-day cycle from cycle 10 to disease progression.
  Arms: MPR+p; MPp+p
Drug: Lenalidomide: Double-blind Maintenance — Single-agent oral lenalidomide 10 mg once daily on Days 1 through 21 of each 28-day cycle from cycle 10 to disease progression.
  Other Names: Revlimid
  Arms: MPR+R
Drug: Lenalidomide: Open-label — Any study participant who had progressive disease had the option of open-label lenalidomide up to 25 mg daily on Days 1 through 21 of each 28-day cycle.
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to determine whether lenalidomide is safe and effective in the treatment of patients with newly diagnosed Multiple Myeloma who are 65 years of age or older.

DETAILED DESCRIPTION:
The three phases for the study as originally defined and as represented in the results of 11 May 2010 are:

Double-blind Treatment Phase: Induction Melphalan/prednisone and lenalidomide 10 mg (MPR) (2 treatment arms), or melphalan/prednisone and placebo (MPp) (1 treatment arm) for up to 9 cycles. If disease progression, subjects have the option to enter into the Open-Label Extension Phase. There is also an option to enter into the Follow-Up Phase. If the disease has not progressed, subject can continue on blinded therapy into Maintenance.

Double-blind Treatment Phase: Maintenance One MPR treatment arm (MPR+R) will continue taking lenalidomide 10 mg in Maintenance. The other MPR treatment arm (MPR+p) will take placebo in Maintenance. The MP p treatment arm will take placebo in Maintenance (MPp+p). If disease progression, subjects have the option to enter the Open-Label Extension Phase to obtain treatment with lenalidomide, or to enter into the Follow-up Phase.

Open-label Extension Phase:

Treatment consists of oral lenalidomide (up to 25 mg) with or without dexamethasone until disease progression or treatment is discontinued for any reason until all study subjects are followed for at least 5 years from the date of randomization or have died. Subjects who discontinue from the Open-Label Extension Phase prior to completing a total of 5 years in the study will enter the Follow-up Phase.

Follow-up Phase:

Subjects are followed for overall survival and subsequent anti-myeloma treatment regimens until all subjects in this study are followed for at least 5 years from randomization or have died.

The pre-planned interim analysis for the Independent Data Monitoring Committee (IDMC) showed that the difference in progression-free survival (PFS) between treatment arms MPR+R and MPp+p (the defined primary comparative analysis for this study) surpassed the pre-specified O'Brien-Fleming boundary for superiority. The IDMC recommended the release of this information to the sponsor and also recommended that all patient and physician study participants receive information concerning the full findings of the MM-015 interim analysis. Therefore, due to these recommendations from the IDMC, treatment-arm codes were sent to the clinical trial centers to unblind the treatment arms of their study subjects once the amended protocol was reviewed and approved by the respective country Health Authorities and Ethics Committees. Subject participation in the MM-015 study continued after unblinding to obtain long-term data for all study endpoints, including overall survival.

When the study was unblinded, subjects still on protocol therapy had completed the Double-Blind Induction, and were on monotherapy in Double-Blind Maintenance. Subjects in arm MPR+R continued their monotherapy on lenalidomide. Subjects in arms MPR+p and MPp+p discontinued their placebo monotherapy and went into an observation period in which no antimyeloma therapy was taken. If disease progressed for any subject, the investigator had the option of entering the subject in Open Label Extension Phase to receive lenalidomide therapy (up to 25 mg daily) or the Follow-up Phase. All subjects were to be followed for at least 5 years from the start of the study.

ELIGIBILITY:
Inclusion Criteria

1. Must understand and voluntarily sign an informed consent form
2. Age greater than or equal to 65 years at the time of signing the informed consent
3. Newly diagnosed with symptomatic multiple myeloma as defined by the 3 criteria below:

MM diagnostic criteria (all of next 3 required)

1. Monoclonal plasma cells in the bone marrow greater than or equal to 10% and/or presence of a biopsy-proven plasmacytoma
2. Monoclonal protein present in the serum and/or urine
3. Myeloma-related organ dysfunction (at least one of the following) [C] Calcium elevation in the blood (serum calcium >10.5mg/dl or upper limit of normal) [R] Renal insufficiency (serum creatinine >2mg/dl) [A] Anemia (hemoglobin <10g/dl or 2g < normal) [B] Lytic bone lesions or osteoporosis AND have measurable disease as defined by the following; IgG multiple myeloma: Serum monoclonal paraprotein (M-protein) level greater than or equal to 1.0 g/dL or urine M-protein level greater than or equal to 200 mg/24 hours IgA multiple myeloma: Serum M-protein level greater than or equal to 0.5 g/dL or urine M-protein level greater than or equal to 200 mg/24 hours IgD multiple myeloma: Serum M-protein level greater than or equal to 0.05 g/dL or urine M-protein level greater than or equal to 200 mg/24 hours Light chain multiple myeloma: Serum M-protein level greater than or equal to 1.0 g/dL or urine M-protein level greater than or equal to 200 mg/24 hours IgM multiple myeloma (IgM M-protein plus lytic bone disease documented by skeletal survey plain films): Serum M-protein level greater than or equal to 1.0g/dL or urine M-protein level greater than or equal to 200mg/24hours
4. Karnofsky performance status greater than or equal to 60%.
5. Able to adhere to the study visit schedule and other protocol requirements.
6. Women of Childbearing potential (WCBP) must:

   a. Have a negative medically supervised pregnancy test prior to the start of study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices and continues sexual abstinence.

   b Either commit to continued abstinence from heterosexual intercourse (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting study drug, during the study therapy (including dose interruptions), and for 28 days after discontinuation of study therapy.
7. Males Subjects must:

   1. Agree to use a condom during sexual contact with a WCBP, even if they have had a vasectomy, throughout study drug therapy, during any dose interruption and after the cessation of study therapy.
   2. Agree to not donate semen during study drug therapy and for a period after end of study drug therapy.
8. All subjects must

   1. Have an understanding that the study drug could have potential teratogenic risk.
   2. Agree to abstain from donating blood while taking study drug therapy and following discontinuation of study drug therapy.
   3. Agree not to share study medication with another person.
   4. All patients must be counseled about pregnancy precautions and risks of fetal exposure.

Female Subjects:

Females of childbearing potential (FCBP) with regular cycles must agree to have pregnancy tests weekly for the first 28 days of study participation and then every 28 days while on study, at study discontinuation, and at day 28 following discontinuation from the study. If menstrual cycles are irregular, the pregnancy testing must occur weekly for the first 28 days and then every 14 days while on study, at study discontinuation, and at days 14 and 28 following discontinuation from the study.

In addition to the required pregnancy testing, the Investigator must confirm with FCBP that she is continuing to use two reliable methods of birth control at each visit. Counseling about pregnancy precautions and the potential risks of fetal exposure must be conducted at a minimum of every 28 days. During counseling, subjects must be reminded to not share study drug and to not donate blood.

Pregnancy testing and counseling must be performed if a subject misses her period or if her pregnancy test or her menstrual bleeding is abnormal. Study drug treatment must be discontinued during this evaluation.

Females must agree to abstain from breastfeeding during study participation and for at least 28 days after the discontinuation from the study.

Male Subjects:

Counseling about the requirement for latex condom use during sexual contact with females of childbearing potential and the potential risks of fetal exposure must be conducted at a minimum of every 28 days. During counseling, subjects must be reminded to not share study drug and to not donate blood, sperm, or semen.

If pregnancy or a positive pregnancy test does occur in a study subject or the partner of a study subject during study participation, study drug must be immediately discontinued.

Exclusion Criteria

1. Previous treatment with antimyeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid [i.e., less than or equal to the equivalent of dexamethasone 40 mg/day for 4 days; such a short course of steroid treatment must not have been given within 28 days [4 weeks] of randomization]).
2. Any serious medical condition, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he or she participates in this study or confounds experimental the ability to interpret data from the study.
3. Pregnant or lactating females.
4. Radiotherapy within 14 days (2 weeks) of randomization.
5. Plasmapheresis within 28 days (4 weeks) of randomization.
6. Any of the following laboratory abnormalities:

   Absolute neutrophil count (ANC) < 1,500 cells/mL (1.5*10^9/L) Platelet count < 75,000 cells/uL (75*10^9/L) for subjects in whom < 50% of bone marrow nucleated cells are plasma cells; but platelet count <30,000/uL for subjects in whom >= 50% of bone marrow nucleated cells are plasma cells Haemoglobin < 8.0 g/dL (80 g/L) Serum creatinine > 2.5 mg/dL (221 µmol/L) Serum aspartate aminotransferase (SGOT/AST) or alanine aminotransferase (SGPT/ALT) > 3.0 times upper limit of normal (ULN)
7. Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for greater than or equal to 3 years.

   Exceptions include the following:

   Basal cell carcinoma of the skin Squamous cell carcinoma of the skin Carcinoma in situ of the cervix Carcinoma in situ of the breast Incidental histologic finding of prostate cancer (TNM Classification of Malignant Tumours (TNM) stage of T1a or T1b)
8. Neuropathy of >= grade 2 severity.
9. Known human immunodeficiency virus (HIV) positivity or active infectious hepatitis, type A, B or C.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 459 (Actual)
Dates: Start 2007-01; Primary Completion 2009-11 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Palumbo, M.D., Principal Investigator — Azienda Sanitaria Ospedaliera Molinette S. Giovanni Battista
Locations (97):
- Australia (8):
  - Hematology Oncology Clinics of Australia, Level 5, Mater Medical Centre, South Brisbane, Queensland
  - Royal Adelaide Hospital Institute of Medical and Veterinary Science, Adelaide, South Australia
  - Royal Prince Alfred Hospital, Camperdown
  - Peter MacCallum Cancer Centre Divsion of Haematology Medical Oncology, East Melbourne
  - Frankston Hospital, Frankston
  - The Alfred Hospital, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
  - Princess Alexandra Hospital, Woolloongabba
- Austria (4):
  - University Hospital Innsbruck, Innsbruck
  - University Hospital of Salzburg St Johanns Spital, Salzburg
  - Medical University of Vienna, Vienna
  - Wilhelminenspital, Vienna
- Belarus (2):
  - Republican Scientific and Practical Centre of Radiation Medicine and Human Ecology, Homyel
  - City Clinical Hospital 9, Minsk
- Belgium (4):
  - AZ St-Jan Brugge Oostende AV, Bruges
  - AZ-VUB, Brussels
  - UZ Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
  - Vseobecna Fakultni Nemocnice v Praze, Prague
- Denmark (2):
  - Hæmatologisk afd. B Aalborg Sygehus Syd, Aalborg
  - Medicinsk afd. Vejle Sygehus, Vejle
- France (5):
  - CHU, Caen
  - CH - Hôpital Dupuytren, Limoges
  - CHU Montpellier- Hopital Lapeyronie, Montpellier
  - Assistance Publique - Hôpitaux de Paris AP-HP, Paris
  - CHU Purpan, Toulouse
- Georgia (2):
  - Ltd M.Zodelava Hematology Centre, Tbilisi
  - Institute of Hematology and Transfusiology, Tbilisi
- Germany (10):
  - Medizinische Klinik und Poliklinik II der Charite Campus Mitte, Berlin
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitatsklinikum Freiburg Medizinische Klinik und Poliklinik, Freiburg im Breisgau
  - Ernst-Moritz-Arndt-Universität Greifswald, Greifswald
  - Universitaetsklinikum Heidelberg Medizinische Klinik und Poliklinik V, Heidelberg
  - Medizinische Klinik und Poliklinik II, Leipzig
  - Poliklinik A, Münster
  - Medizinische Klinik - Abteilung II, Tübingen
  - Medizinische Universitatsklinik, Ulm
  - Medizinische Klinik und Poliklinik II des Universitatsklinikums Wurzburg, Würzburg
- Greece (3):
  - G. GENNIMATAS General Hospital of Athens Department of Hematolgosy, Athens
  - General Air Force Hospital, Athens
  - Alexandra General Hospital of Athens, Athens
- Ireland (2):
  - Hope Directorate Haematology Oncology Service St. James Hospital, Dublin
  - Midlands Regional, Tullamore / Co Offally
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Hematology Institute, Hemato-Oncology Division,Davidoff Cancer Center, Rabin MC Beilinson Hospital, Petch Tikva
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (8):
  - Policlinico S. Orsola, Bologna
  - A.O.U. San Martino, Genova
  - Dipartmento Oncologico Struttura Complessa di ematlologiaA.O. Ospedale Niguarda Ca Granda, Milan
  - Policlinico San Matteo Universita Di Pavia, Pavia
  - Divisione Di Ematologia Ospedale Cattedra di Ematologia, Rome
  - Azienda Policlinico Umberto I, Universita La Sapienzadi Roma, Rome
  - Dipartimento di Onco-Ematologia, San Giovanni Rotondo (FG)
  - Azienda Sanitaria Ospedaliera Molinette S. Giovanni Battista, Turin
- Netherlands (4):
  - VU Medical Center, Amsterdam
  - Erasmus Medical Center, Rotterdam
  - Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (6):
  - Klinika Hematologii Samodzielny Publiczny Szpital Kliniczny Akademii, Bialystok
  - Institute of Internal Diseases University of Medicine, Gdansk
  - Oddzial Kliniczny Kliniki Hematologii, Krakow
  - Uniwersytet Medyczny w Lodzi, Lodz
  - University School of Medicine, Lublin
  - Akademia Medyczna w Warszawie Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- Russia (7):
  - Burdenko Central Military Clinical Hospital, Moscow
  - Institution of Russian Academy of Medical Sciences Russian Oncological Research Centre n.a. N. N. Bl, Moscow
  - Moscow Regional Research Institute n.a. Vladimirsky, Moscow
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Medical Radiological Research Center RAMS, Obninsk
  - St. Petersburg Research Institute of Hematology and Blood Transfusion, Saint Petersburg
  - Samara Regional Clinical Hospital, Samara
- Spain (5):
  - Hospital Clinic, Barcelona
  - Hospital Universitaro Puerta del MarServicio de Hematologia, Cadiz
  - Hospital Universitario de la Princessa, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Virgen del Rocio Servicio de Hematologia, Seville
- Sweden (2):
  - Medicinkliniken, Borås
  - Medicinska kliniken, Malmo
- UniversitatsSpital ZurichKlinik fur Onkologie, Zurich, Switzerland
- Turkey (Türkiye) (3):
  - Ankara University, Ankara
  - Marmara School of Medicine, Istanbul
  - Ege University Medical School, Izmir
- Ukraine (6):
  - Cherkassy Regional Oncology Center, Cherkassy
  - Dnepropetrovsk City Clinical Hospital 4, Dnipro
  - Institute of Urgent and Recovery Surgery, Donetsk
  - Institute of Hematology and Transfusiology of the UAMS Department of blood diseases, Kiev
  - Institute of Blood Pathology and Transfusion Medicine of the AMS of Ukraine, Lviv
  - Zhitomir Regional Clinical Hospital, Zhytomyr
- United Kingdom (5):
  - Monklands Hospital, Aidrie
  - St James's University Hospital, Leeds
  - University College London Hospitals Cancer Clinical Trials Unitist FloorCentral wing, London
  - Kings College Hospital, London
  - Christie NHS Trust Hospital, Manchester

REFERENCES:
- [Result] Dimopoulos MA, Delforge M, Hajek R, Kropff M, Petrucci MT, Lewis P, Nixon A, Zhang J, Mei J, Palumbo A. Lenalidomide, melphalan, and prednisone, followed by lenalidomide maintenance, improves health-related quality of life in newly diagnosed multiple myeloma patients aged 65 years or older: results of a randomized phase III trial. Haematologica. 2013 May;98(5):784-8. doi: 10.3324/haematol.2012.074534. Epub 2012 Dec 14. PMID 23242595
- [Result] Palumbo A, Hajek R, Delforge M, Kropff M, Petrucci MT, Catalano J, Gisslinger H, Wiktor-Jedrzejczak W, Zodelava M, Weisel K, Cascavilla N, Iosava G, Cavo M, Kloczko J, Blade J, Beksac M, Spicka I, Plesner T, Radke J, Langer C, Ben Yehuda D, Corso A, Herbein L, Yu Z, Mei J, Jacques C, Dimopoulos MA; MM-015 Investigators. Continuous lenalidomide treatment for newly diagnosed multiple myeloma. N Engl J Med. 2012 May 10;366(19):1759-69. doi: 10.1056/NEJMoa1112704. PMID 22571200
- [Derived] Dimopoulos MA, Petrucci MT, Foa R, Catalano J, Kropff M, Terpos E, Zhang J, Grote L, Jacques C, Palumbo A; MM-015 Investigators. Impact of maintenance therapy on subsequent treatment in patients with newly diagnosed multiple myeloma: use of "progression-free survival 2" as a clinical trial end-point. Haematologica. 2015 Aug;100(8):e328-30. doi: 10.3324/haematol.2014.120790. Epub 2015 Apr 3. No abstract available. PMID 25840600

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data represents a May 11, 2010 data cut-off. The study is ongoing.
Pre-assignment Details: Of the 606 subjects screened for this study, 147 failed screening. Reasons for screen failures included: laboratory values not met (45 subjects); diagnostic criteria for measurable multiple myeloma not met (30 subjects); other inclusion/exclusion criteria not met (30 subjects); subject withdrawal of consent (14 subjects); and other (28 subjects).
Period: Double-blind Treatment
Arm/Group | MPR+R | MPR+p | MPp+p
Started | 152 (Intent to treat population of all randomized participants) | 153 | 154
Safety Population | 150 (Participants who took at least one dose of study drug.) | 152 | 153
Completed | 0 (Double-blind Treatment Period had no defined completion.) | 0 | 0
Not Completed | 152 | 153 | 154
Not completed — Ongoing in Double-blind Treatment | 45 | 24 | 18
Not completed — Adverse Event | 31 | 27 | 12
Not completed — Disease Progression | 47 | 81 | 102
Not completed — Lack of Efficacy | 1 | 4 | 2
Not completed — Withdrawal by Subject | 15 | 9 | 10
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 4 | 4 | 4
Not completed — Protocol Violation | 1 | 0 | 2
Not completed — Other | 7 | 4 | 4
Period: Open-label Extension
Arm/Group | MPR+R | MPR+p | MPp+p
Started | 19 | 47 | 72
Completed | 0 (Participants continue until disease progression or other reason for discontinuing.) | 0 | 0
Not Completed | 19 | 47 | 72
Not completed — Ongoing in Open Label Period | 7 | 15 | 25
Not completed — Adverse Event | 1 | 3 | 7
Not completed — Disease Progression | 8 | 23 | 26
Not completed — Withdrawal by Subject | 2 | 3 | 3
Not completed — Death | 1 | 2 | 4
Not completed — Other | 0 | 1 | 7
Period: Follow-up
Arm/Group | MPR+R | MPR+p | MPp+p
Started | 75 (66 participants from Double-blind and 9 from the Open Label Extension) | 90 (65 participants from the Double-blind and 25 from the Open Label Extension) | 88 (52 participants from the Double-blind and 36 from the Open Label Extension)
Completed | 0 | 0 | 0
Not Completed | 75 | 90 | 88
Not completed — Ongoing in Follow-up Period | 52 | 51 | 60
Not completed — Death | 21 | 31 | 24
Not completed — Lost to Follow-up | 2 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MPR+R | MPR+p | MPp+p | Total
Number analyzed (Participants) | 152 | 153 | 154 | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (5.33) | 72.1 (5.20) | 72.0 (5.26) | 72.0 (5.25)
Age, Customized [Number; unit: participants]
  <=75 years | 116 | 116 | 116 | 348
  >75 years | 36 | 37 | 38 | 111
Gender [Count of Participants; unit: Participants]
  Female | 81 | 71 | 79 | 231
  Male | 71 | 82 | 75 | 228
Race/Ethnicity, Customized [Number; unit: participants]
  White | 151 | 151 | 151 | 453
  Black | 1 | 0 | 0 | 1
  Hispanic | 0 | 0 | 1 | 1
  Asian / Pacific Islander | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Other | 0 | 2 | 2 | 4
Weight [Mean (Standard Deviation); unit: kilograms] | 73.5 (14.77) | 72.0 (12.79) | 72.1 (15.20) | 72.5 (14.28)
Height [Mean (Standard Deviation); unit: centimeter] | 164.8 (9.81) | 165.3 (9.33) | 165.7 (9.79) | 165.3 (9.63)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 133.9 (17.71) | 135.5 (18.60) | 136.4 (20.13) | 135.3 (18.83)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78.5 (9.53) | 77.4 (9.99) | 78.8 (10.40) | 78.2 (9.98)
Temperature [Mean (Standard Deviation); unit: degrees centigrade] | 36.5 (0.41) | 36.5 (0.38) | 36.5 (0.40) | 36.5 (0.40)
Pulse [Mean (Standard Deviation); unit: beats per minute] | 76.0 (9.77) | 77.3 (10.50) | 76.3 (10.80) | 76.5 (10.36)
Karnofsky Performance Scale [Mean (Standard Deviation); unit: units on a scale] — Karnofsky Performance Scale classifies patients according to their functional impairment. Scores range from 0-100, the lower the score, the greater the impairment and worse prospect of survival for most serious illnesses.
  units on a scale | 81.1 (11.95) | 82.2 (11.71) | 84.0 (11.46) | 82.4 (11.74)
International Staging System (ISS) [Number; unit: participants] — ISS form multiple myeloma divides myeloma into 3 stages based only on the serum beta-2 microglobulin and serum albumin levels. Higher stages represent more advanced disease.
  participants
    Stage I | 28 | 32 | 28 | 88
    Stage II | 50 | 47 | 48 | 145
    Stage III | 74 | 74 | 78 | 226
Creatinine clearance [Number; unit: participants]
  >=60 ml/min | 72 | 83 | 77 | 232
  <60 ml/min | 78 | 69 | 76 | 223
  Missing | 2 | 1 | 1 | 4
Beta2 Microglobulin [Number; unit: participants]
  >5.5 mg/L | 74 | 78 | 67 | 219
  <=5.5 mg/L | 77 | 75 | 87 | 239
  Missing | 1 | 0 | 0 | 1
Albumin [Number; unit: participants]
  >35 g/L | 87 | 82 | 81 | 250
  <= 35 g/L | 63 | 70 | 72 | 205
  Missing | 2 | 1 | 1 | 4
C-reactive Protein [Number; unit: participants]
  >4 mg/L | 65 | 56 | 64 | 185
  <=4 mg/L | 84 | 94 | 89 | 267
  Missing | 3 | 3 | 1 | 7
Multiple Myeloma Subtype [Number; unit: participants]
  Immunoglobulin A (IgA) | 39 | 38 | 33 | 110
  Other | 108 | 112 | 116 | 336
  Missing | 5 | 3 | 5 | 13
Plasma Cells in the Bone Marrow [Mean (Standard Deviation); unit: percentage of plasma cells] | 39.8 (24.79) | 39.3 (25.01) | 37.9 (23.65) | 39.0 (24.45)

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimates of Progression-free Survival (PFS) Based on the Response Assessment by the Central Adjudication Committee (CAC)
Description: Data as of 11 May 2010 cutoff. PFS was calculated as the time from randomization to the earlier of the first documentation of progressive disease (PD) as determined by the CAC, or death on study due to any cause. PD was based on the European Group for Blood and Marrow Transplantation/International Bone Marrow Transplant Registry/Autologous Bone Marrow Transplant Registry [EBMT/IBMTR/ABMTR] criteria.
  PD criteria includes increasing monoclonal paraprotein levels, bone marrow findings, worsening lytic bone disease, progressively enlarging extramedullary plasmacytomas, or hypercalcemia.
Time Frame: up to 165 weeks
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
weeks | 136.1 [86.14 to NA] — Upper limit not estimable because of the number of participants without progressive disease at data cut-off. | 62.1 [56.14 to 72.14] | 56.1 [52.14 to 68.14]
Statistical Analysis 1: Comparison: MPR+R vs MPp+p; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value is based on unstratified log rank test of Kaplan-Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.395, 95% CI 2-sided [0.278 to 0.560]
Statistical Analysis 2: Comparison: MPR+R vs MPR+p; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value is based on unstratified log rank test of Kaplan-Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.494, 95% CI 2-sided [0.347 to 0.702]
Statistical Analysis 3: Comparison: MPR+p vs MPp+p; Test type: Superiority or Other; p = 0.134, Log Rank — The p-value is based on unstratified log rank test of Kaplan-Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.796, 95% CI 2-sided [0.589 to 1.075]

2. Secondary Outcome: Kaplan Meier Estimates of Progression-free Survival (PFS) From Start of Maintenance Therapy Period Based on the Response Assessment by the Central Adjudication Committee (CAC)
Description: Data as of 11 May 2010 cutoff. PFS calculated from the start of the Maintenance period to the earlier of the first documentation of progressive disease (PD) as determined by the CAC, or death on study due to any cause.
  PD was based on the European Group for Blood and Marrow Transplantation/International Bone Marrow Transplant Registry/Autologous Bone Marrow Transplant Registry [EBMT/IBMTR/ABMTR] criteria.
  PD criteria includes increasing monoclonal paraprotein levels, bone marrow findings, worsening lytic bone disease, progressively enlarging extramedullary plasmacytomas, or hypercalcemia.
Time Frame: Approximately week 37 (start of cycle 10) to week 165
Population: Intent to treat (ITT) population of participants in Arms MPR+R and MPR+p who entered maintenance within the Double-blind Treatment Period
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MPR+R | MPR+p
Number analyzed (Participants) | 88 | 94
weeks | 112.0 [83.29 to NA] — Upper limit not estimable because of the number of participants without progressive disease at data cut-off. | 32.3 [23.57 to 52.14]
Statistical Analysis 1: Comparison: MPR+R vs MPR+p; Test type: Superiority or Other; p < 0.001, Log Rank; P-value is based on unstratified log rank test of Kaplan-Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.340, 95% CI 2-sided [0.214 to 0.541]

3. Secondary Outcome: Kaplan Meier Estimates of Overall Survival (OS)
Description: Data as of 11 May 2010 cutoff. Overall survival (OS) was defined as the time between randomization and death. Participants who died, regardless of the cause of death, were considered to have had an event. Participants who were lost to follow-up prior to the end of the trial, or who were withdrawn from the trial, were censored at the time of last contact. Participants who were still being treated were censored at the last available date available, or clinical cut-off date, if it was earlier.
Time Frame: up to 177 weeks
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
weeks | NA [NA to NA] — Not able to estimate since few participants died as of the May 11, 2010 cut-off. | NA [148.43 to NA] — Not able to estimate since few participants died as of the May 11, 2010 cut-off. | NA [NA to NA] — Not able to estimate since few participants died as of the May 11, 2010 cut-off.

4. Secondary Outcome: Kaplan Meier Estimates of Time to Progression (TTP) Based on the Response Assessment by the Central Adjudication Committee (CAC)
Description: Data as of 11 May 2010 cutoff. TTP was the time between randomization and disease progression as determined by the CAC. PD was based on the European Group for Blood and Marrow Transplantation/International Bone Marrow Transplant Registry/Autologous Bone Marrow Transplant Registry [EBMT/IBMTR/ABMTR] criteria.
  PD criteria includes increasing monoclonal paraprotein levels, bone marrow findings, worsening lytic bone disease, progressively enlarging extramedullary plasmacytomas, or hypercalcemia.
Time Frame: up to 165 weeks
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
weeks | 148.1 [100.00 to NA] — Upper limit not estimable because of the number of participants without progressive disease at data cut-off. | 62.7 [57.14 to 74.14] | 61.3 [52.29 to 70.14]
Statistical Analysis 1: Comparison: MPR+R vs MPp+p; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value is based on unstratified log rank test of Kaplan-Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.337, 95% CI 2-sided [0.231 to 0.493]
Statistical Analysis 2: Comparison: MPR+R vs MPR+p; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value is based on unstratified log rank test of Kaplan-Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.414, 95% CI 2-sided [0.284 to 0.603]
Statistical Analysis 3: Comparison: MPR+p vs MPp+p; Test type: Superiority or Other; p = 0.223, Log Rank — The p-value is based on unstratified log rank test of Kaplan-Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.826, 95% CI 2-sided [0.606 to 1.125]

5. Secondary Outcome: Number of Participants in Disease Response Categories Representing Their Best Response During the Double-blind Treatment Period
Description: Data as of 11 May 2010 cutoff. Best response was determined by the Central Assessment Committee (CAC) based on the European Group for Blood and Marrow Transplantation (EBMT) criteria: Complete Response (CR)-absence of serum and urine monoclonal paraprotein for 6 weeks, plus no increase in size or number of bone lesions, plus other factors); Partial Response (PR)-not all CR criteria, plus >=50% reduction in serum monoclonal paraprotein plus others; Stable Disease (SD)- not PR or PD; Progressive Disease (PD)- reappearance of monoclonal paraprotein, bone lesions, other; Not Evaluable (NE).
Time Frame: Up to 165 weeks
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
participants
  Complete response (CR) | 15 | 5 | 5
  Partial response (PR) | 102 | 99 | 72
  Stable disease (SD) | 28 | 40 | 70
  Progressive disease (PD) | 0 | 2 | 0
  Response not evaluable (NE) | 7 | 7 | 7
Statistical Analysis 1: Comparison: MPR+R vs MPp+p; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value calculation excludes the category - Response not evaluable (NE)
Statistical Analysis 2: Comparison: MPR+R vs MPR+p; Test type: Superiority or Other; p = 0.009, Wilcoxon (Mann-Whitney) — P-value calculation excludes the category - Response not evaluable (NE)
Statistical Analysis 3: Comparison: MPR+p vs MPp+p; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney) — P-value calculation excludes the category - Response not evaluable (NE)
Statistical Analysis 4: Comparison: MPR+R vs MPp+p; Based on dichotomized response: 1) CR or PR 2) SD or PD or NE; Test type: Superiority or Other; p < 0.001, Fisher Exact; Odds Ratio (OR) = 3.34, 95% CI 2-sided [2.04 to 5.47]
Statistical Analysis 5: Comparison: MPR+R vs MPR+p; Based on dichotomized response: 1) CR or PR 2) SD or PD or NE; Test type: Superiority or Other; p = 0.096, Fisher Exact; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.95 to 2.62]
Statistical Analysis 6: Comparison: MPR+p vs MPp+p; Based on dichotomized response: 1) CR or PR 2) SD or PD or NE; Test type: Superiority or Other; p = 0.002, Fisher Exact; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.33 to 3.37]

6. Secondary Outcome: Time to First Response
Description: Data as of 11 May 2010 cutoff. Time to first response was defined as the time from start of treatment until first response as assessed by the Central Assessment Committee (CMC) based on European Group for Blood and Marrow Transplantation (EBMT) criteria.
Time Frame: Up to 66 weeks
Population: Participants who had a partial response (PR) or complete response (CR)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 117 | 104 | 77
weeks | 10.0 (7.40) | 9.3 (6.55) | 16.2 (11.59)

7. Secondary Outcome: Kaplan Meier Estimates for Duration of Response as Determined by the Central Adjudication Committee (CAC)
Description: Data as of 11 May 2010 cutoff. Duration of myeloma response was defined as the time from the initial response date to the earlier of progressive disease (PD) as determined by the CAC or death on study. PD was based on the European Group for Blood and Marrow Transplantation/International Bone Marrow Transplant Registry/Autologous Bone Marrow Transplant Registry [EBMT/IBMTR/ABMTR] criteria.
  PD criteria includes increasing monoclonal paraprotein levels, bone marrow findings, worsening lytic bone disease, progressively enlarging extramedullary plasmacytomas, or hypercalcemia.
Time Frame: Up to 149 weeks
Population: Population: Participants who achieved a partial response (PR) or complete response (CR).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 117 | 104 | 77
weeks | 121.6 [96.00 to NA] — Upper limit not estimable because of the number of participants without progressive disease at data cut-off. | 56.1 [52.14 to 64.29] | 55.4 [44.14 to 76.14]
Statistical Analysis 1: Comparison: MPR+R vs MPp+p; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value is based on unstratified log rank test of Kaplan Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.348, 95% CI 2-sided [0.228 to 0.531]
Statistical Analysis 2: Comparison: MPR+R vs MPR+p; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value is based on unstratified log rank test of Kaplan Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.419, 95% CI 2-sided [0.281 to 0.623]
Statistical Analysis 3: Comparison: MPR+p vs MPp+p; Test type: Superiority or Other; p = 0.302, Log Rank — The p-value is based on unstratified log rank test of Kaplan Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.825, 95% CI 2-sided [0.571 to 1.191]

8. Secondary Outcome: Kaplan Meier Estimates for Time to Next Antimyeloma Therapy
Description: Data as of 11 May 2010 cutoff. Time to the next antimyeloma therapy was defined as time from randomization to the start of another non-protocol antimyeloma therapy. Participants who do not receive another anti-myeloma therapy were censored at the last assessment or follow-up visit known to have received no new therapy.
Time Frame: Up to 168 weeks
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
weeks | 128.9 [99.86 to NA] — Upper limit not estimable because of the number of participants who had not started a non-protocol anti-myeloma therapy at data cut-off. | 66.1 [60.14 to 76.00] | 66.3 [61.14 to 72.43]
Statistical Analysis 1: Comparison: MPR+R vs MPp+p; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value is based on unstratified log rank test of Kaplan Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.404, 95% CI 2-sided [0.296 to 0.553]
Statistical Analysis 2: Comparison: MPR+R vs MPR+p; Test type: Superiority or Other; p < 0.001, Log Rank — The p-value is based on unstratified log rank test of Kaplan Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.499, 95% CI 2-sided [0.363 to 0.688]
Statistical Analysis 3: Comparison: MPR+p vs MPp+p; Test type: Superiority or Other; p = 0.169, Log Rank — The p-value is based on unstratified log rank test of Kaplan Meier curve differences between the treatment groups; Hazard Ratio (HR) = 0.827, 95% CI 2-sided [0.630 to 1.085]

9. Secondary Outcome: Summary of Participants With Treatment-Emergent Adverse Events (TEAE) During the Double-Blind Treatment Period
Description: Data as of 11 May 2010 cutoff. Participant counts in different categories of TEAEs during the double-blind treatment period. A TEAE is as any AE occurring or worsening on or after the first treatment of any study drug, and within 30 days after the last dose of the last study drug. Severity grades according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE) on a 1-5 scale: Grade 1= Mild AE, Grade 2= Moderate AE, Grade 3= Severe AE, Grade 4= Life-threatening or disabling AE, Grade 5=Death related to AE. Dose reduction includes reduction with or without interruption.
Time Frame: Up to 169 weeks (Double-blind therapy period plus 4 weeks)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 150 | 152 | 153
participants
  >=1 adverse event (AE) | 150 | 151 | 153
  >=1 CTCAE grade 3-4 AE | 137 | 129 | 107
  >=1 CTCAE grade 5 AE | 7 | 6 | 7
  >=1 serious AE (SAE) | 66 | 62 | 56
  >=1 AE related to Lenaldomide/Placebo | 148 | 145 | 131
  >=1 AE related to Melphalan | 140 | 134 | 126
  >=1AE related to Prednisone | 87 | 94 | 93
  >=1 Grade 3-4 AE related to Lenaldomide/Placebo | 128 | 117 | 68
  >=1 Grade 3-4 AE related to Melphalan | 118 | 110 | 62
  >=1 Grade 3-4 AE related to Prednisone | 32 | 29 | 22
  >=1 Grade 5 AE related to Lenalidomide/Placebo | 3 | 2 | 2
  >=1 Grade 5 AE related to Melphalan | 3 | 1 | 3
  >=1 Grade 5 AE related to Prednisone | 1 | 1 | 1
  >=1 SAE related to Lenalidomide/Placebo | 38 | 32 | 11
  >=1 SAE related to Melphalan | 27 | 24 | 11
  >=1 SAE related to Prednisone | 19 | 16 | 5
  >=1 AE leading to Lenalidomide/Placebo withdrawal | 26 | 24 | 14
  >=1 AE leading to Melphalan withdrawal | 20 | 19 | 10
  >=1 AE leading to Prednisone withdrawal | 20 | 19 | 10
  >=1 AE leading to Lenalidomide/Plac dose reduction | 71 | 70 | 26
  >=1 AE leading to Melphalan dose reduction | 47 | 58 | 21
  >=1 AE leading to Prednisone dose reduction | 15 | 7 | 5
  >=1 AE leading to Lenalidomide/Plac dose interrupt | 92 | 82 | 51
  >=1 AE leading to Melphalan dose interruption | 5 | 1 | 0
  >=1 AE leading to Prednisone dose interruption | 28 | 39 | 15

10. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Global Quality of Life Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLC-C30 is a 30-item questionnaire to assess the quality of life in cancer patients. EORTC QLQ-C30 includes functional scales (physical, role, cognitive, emotional, social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnoea, appetite loss, insomnia, constipation/diarrhea, financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); two used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score = better quality of life.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=114,121,125) | 2.3 (26.13) | 5.6 (18.86) | 6.1 (19.41)
  Cycle 7 - approximately Month 7 (n=96,108,110) | 8.0 (24.95) | 8.1 (22.48) | 4.2 (23.92)
  Cycle 10 - approximately Month 10 (n=84,86,96) | 12.4 (25.33) | 8.8 (24.70) | 6.2 (24.60)
  Cycle 13 - approximately Month 13 (n=70,70,82) | 7.6 (28.32) | 8.8 (24.02) | 5.4 (22.80)
  Cycle 16 - approximately Month 16 (n=61,50,62) | 10.7 (25.28) | 7.2 (26.29) | 8.1 (25.11)

11. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Physical Functioning Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score=better level of physical functioning.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=120,127,130) | 1.9 (23.72) | 3.3 (21.64) | 4.5 (18.68)
  Cycle 7 - approximately Month 7 (n=100,112,112) | 8.2 (22.71) | 8.1 (20.54) | 2.7 (23.20)
  Cycle 10 - approximately Month 10 (n=88,95,96) | 8.9 (22.75) | 8.5 (25.62) | 5.1 (20.42)
  Cycle 13 - approximately Month 13 (n=75,74,83) | 8.6 (24.04) | 9.7 (25.39) | 3.3 (20.30)
  Cycle 16 - approximately Month 16 (n=64,53,63) | 10.0 (25.00) | 7.6 (22.66) | 1.1 (19.30)

12. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Role Functioning Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score=better level of role functioning.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=119,127,130) | 1.8 (33.18) | 3.0 (30.75) | 7.4 (26.34)
  Cycle 7 - approximately Month 7 (n=99,112,113) | 5.7 (35.57) | 8.0 (32.42) | 6.9 (31.16)
  Cycle 10 - approximately Month 10 (n=86,95,95) | 9.3 (35.76) | 7.5 (36.29) | 5.6 (31.29)
  Cycle 13 - approximately Month 13 (n=74,74,82) | 9.7 (40.36) | 11.7 (33.42) | 5.7 (30.68)
  Cycle 16 - approximately Month 16 (n=64,53,63) | 12.2 (40.09) | 8.5 (34.22) | 7.1 (31.93)

13. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Emotional Functioning Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score = better level of emotional functioning.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=115,125,128) | 4.8 (25.00) | 2.7 (22.59) | 6.8 (18.75)
  Cycle 7 - approximately Month 7 (n=98,111,112) | 8.8 (24.94) | 4.2 (20.38) | 5.0 (21.56)
  Cycle 10 - approximately Month 10 (n=86,92,97) | 9.0 (23.28) | 1.6 (22.07) | 4.7 (22.05)
  Cycle 13 - approximately Month 13 (n=73,73,83) | 8.2 (24.59) | 1.1 (21.78) | 6.6 (21.78)
  Cycle 16 - approximately Month 16 (n=63,52,63) | 9.9 (23.23) | -0.2 (21.57) | 6.9 (19.72)

14. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Congitive Functioning Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score = better level of cognitive functioning.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=115,125,128) | 0.3 (21.51) | -2.0 (21.33) | 1.3 (16.68)
  Cycle 7 - approximately Month 7 (n=98,111,113) | 2.9 (22.31) | 0.1 (17.33) | 0.7 (18.42)
  Cycle 10 - approximately Month 10 (n=87,92,97) | 1.0 (22.64) | -4.4 (19.89) | -2.7 (20.65)
  Cycle 13 - approximately Month 13 (n=73,73,83) | -0.0 (21.34) | -3.0 (23.78) | -1.4 (17.69)
  Cycle 16 - approximately Month 16 (n=63,52,63) | 0.3 (22.29) | -3.5 (27.48) | -4.0 (18.13)

15. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Social Functioning Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score = better level of social functioning.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=115,125,127) | 5.1 (35.05) | 0.3 (26.60) | 6.0 (22.78)
  Cycle 7 - approximately Month 7 (n=98,111,112) | 8.3 (33.87) | 4.4 (24.48) | 6.1 (26.57)
  Cycle 10 - approximately Month 10 (n=87,92,97) | 10.9 (34.27) | 4.5 (29.87) | 4.1 (27.22)
  Cycle 13 - approximately Month 13 (n=72,73,83) | 11.8 (32.91) | 7.5 (29.80) | 6.2 (27.63)
  Cycle 16 - approximately Month 16 (n=63,52,63) | 13.2 (33.35) | 6.1 (30.79) | 9.8 (28.66)

16. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Fatigue Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the fatigue scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=120,127,129) | -3.0 (25.61) | -5.5 (24.08) | -5.1 (24.33)
  Cycle 7 - approximately Month 7 (n=100,112,110) | -7.6 (23.00) | -9.5 (25.97) | -5.7 (27.32)
  Cycle 10 - approximately Month 10 (n=87,95,95) | -7.5 (27.31) | -7.5 (29.78) | -6.9 (28.31)
  Cycle 13 - approximately Month 13 (n=74,74,82) | -7.1 (26.08) | -10.7 (30.33) | -7.5 (27.29)
  Cycle 16 - approximately Month 16 (n=64,53,62) | -10.0 (26.86) | -9.7 (28.77) | -4.1 (26.34)

17. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Nausea and Vomiting Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the nausea/vomiting scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=120,127,130) | 3.3 (19.40) | -1.3 (17.14) | -0.0 (17.36)
  Cycle 7 - approximately Month 7 (n=99,112,112) | 0.5 (14.57) | -0.7 (19.94) | 0.7 (14.73)
  Cycle 10 - approximately Month 10 (n=87,95,97) | 1.9 (16.75) | -1.4 (19.40) | 0.3 (14.23)
  Cycle 13 - approximately Month 13 (n=75,72,83) | 0.7 (13.55) | -3.0 (19.65) | -0.4 (12.48)
  Cycle 16 - approximately Month 16 (n=64,52,62) | 1.0 (12.90) | -4.2 (18.65) | -1.3 (9.21)

18. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Pain Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the pain scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=120,127,129) | -14.4 (32.76) | -13.8 (33.60) | -13.4 (29.32)
  Cycle 7 - approximately Month 7 (n=100,112,113) | -17.8 (36.18) | -16.5 (33.45) | -11.5 (33.49)
  Cycle 10 - approximately Month 10 (n=88,95,97) | -17.2 (34.78) | -15.6 (35.30) | -9.8 (31.71)
  Cycle 13 - approximately Month 13 (n=74,74,83) | -13.7 (40.48) | -14.9 (33.28) | -12.1 (27.46)
  Cycle 16 - approximately Month 16 (n=64,53,63) | -20.3 (33.92) | -11.0 (33.00) | -12.2 (29.96)

19. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Dyspnoea Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the dyspnoea scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=117,126,126) | -2.6 (29.74) | -6.4 (32.04) | -0.0 (23.48)
  Cycle 7 - approximately Month 7 (n=100,110,110) | -1.7 (28.18) | -8.5 (32.07) | 2.1 (20.82)
  Cycle 10 - approximately Month 10 (n=86,93,96) | -4.3 (30.60) | -4.3 (35.87) | 3.8 (25.07)
  Cycle 13 - approximately Month 13 (n=73,73,81) | -5.0 (30.26) | -2.3 (30.60) | -0.0 (22.35)
  Cycle 16 - approximately Month 16 (n=62,53,62) | -3.2 (29.39) | -6.3 (32.07) | 1.6 (22.92)

20. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Insomnia Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the insomnia scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=118,124,128) | 2.0 (33.56) | -1.6 (31.77) | -5.0 (27.77)
  Cycle 7 - approximately Month 7 (n=100,109,111) | -1.0 (29.76) | -6.4 (27.02) | -5.7 (32.06)
  Cycle 10 - approximately Month 10 (n=87,94,96) | -5.0 (28.99) | -2.5 (25.04) | -1.7 (32.58)
  Cycle 13 - approximately Month 13 (n=75,73,83) | -4.9 (29.86) | 0.9 (29.38) | -6.8 (29.80)
  Cycle 16 - approximately Month 16 (n=64,53,63) | -4.7 (32.46) | -0.6 (32.36) | -3.7 (31.18)

21. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Appetite Loss Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the appetite loss scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=119,125,130) | 1.7 (36.54) | 1.9 (34.73) | -5.6 (25.96)
  Cycle 7 - approximately Month 7 (n=99,111,111) | -3.7 (33.64) | -5.7 (31.75) | -5.7 (27.66)
  Cycle 10 - approximately Month 10 (n=87,93,96) | -5.0 (33.15) | -5.4 (29.20) | -8.0 (29.32)
  Cycle 13 - approximately Month 13 (n=75,72,83) | -6.2 (36.23) | -8.8 (30.13) | -4.8 (32.15)
  Cycle 16 - approximately Month 16 (n=64,52,63) | -7.8 (36.01) | -16.0 (35.24) | -6.4 (28.62)

22. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Constipation Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the constipation scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=114,124,128) | -1.8 (34.31) | 4.8 (30.86) | -4.9 (27.45)
  Cycle 7 - approximately Month 7 (n=96,111,112) | -3.5 (36.35) | 0.6 (30.14) | -2.7 (31.05)
  Cycle 10 - approximately Month 10 (n=86,93,97) | -5.0 (34.88) | -1.1 (28.43) | -1.7 (26.95)
  Cycle 13 - approximately Month 13 (n=73,73,81) | -5.0 (31.27) | -2.7 (28.74) | -3.3 (29.16)
  Cycle 16 - approximately Month 16 (n=63,51,62) | -1.6 (31.36) | -5.2 (30.82) | -2.2 (32.44)

23. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Diarrhoea Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the diarrhea scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=115,125,124) | 2.3 (28.85) | 1.9 (24.06) | 3.2 (25.65)
  Cycle 7 - approximately Month 7 (n=98,109,112) | 3.4 (25.54) | -1.2 (23.09) | 0.9 (22.13)
  Cycle 10 - approximately Month 10 (n=87,92,95) | 1.1 (22.98) | 1.4 (20.91) | -0.0 (21.19)
  Cycle 13 - approximately Month 13 (n=73,73,80) | 5.5 (30.43) | -1.4 (18.78) | 0.8 (18.35)
  Cycle 16 - approximately Month 16 (n=63,52,61) | 10.6 (35.83) | 1.3 (19.75) | 0.5 (17.74)

24. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13 and 16 in European Organization for Research and Treatment of Cancer Questionnaire for Patients With Cancer (EORTC QLQ-C30) Financial Difficulties Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a problem scale like the financial problems scale = higher level of financial problems.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=111,123,125) | 2.4 (24.91) | -1.1 (19.06) | -2.9 (18.93)
  Cycle 7 - approximately Month 7 (n=94,111,112) | 2.1 (23.85) | -0.6 (28.07) | -2.1 (22.50)
  Cycle 10 - approximately Month 10 (n=84,92,97) | 6.0 (21.44) | 0.7 (28.81) | -1.7 (19.47)
  Cycle 13 - approximately Month 13 (n=70,72,83) | 4.8 (21.45) | -0.5 (28.80) | -4.0 (26.75)
  Cycle 16 - approximately Month 16 (n=61,52,63) | 1.6 (20.58) | -0.6 (35.24) | -5.3 (30.06)

25. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13, 16 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Disease Symptoms Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. EORTC QLQ-MY20 includes four scales: disease symptoms, treatment side-effects, future perspective, and body image. Questions used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale; higher score for the disease symptoms scale = higher level of symptomatology.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=113,121,127) | -8.9 (19.56) | -8.7 (19.13) | -5.4 (15.83)
  Cycle 7 - approximately Month 7 (n=96,109,112) | -9.0 (20.64) | -9.7 (23.25) | -6.0 (20.81)
  Cycle 10 - approximately Month 10 (n=85,91,95) | -7.9 (23.00) | -7.1 (23.85) | -5.4 (18.79)
  Cycle 13 - approximately Month 13 (n=72,73,82) | -7.2 (25.91) | -8.8 (24.90) | -6.3 (21.84)
  Cycle 16 - approximately Month 16 (n=62,51,62) | -10.5 (23.87) | -5.9 (25.79) | -3.3 (20.67)

26. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13, 16 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) In Side Effects of Treatment Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. Questions used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale; higher score for the side effects scale = higher level of symptomatology.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=113,120,125) | 1.3 (13.37) | 0.1 (13.28) | 0.6 (12.67)
  Cycle 7 - approximately Month 7 (n=95,108,111) | 0.4 (15.22) | -1.7 (14.27) | 1.8 (12.94)
  Cycle 10 - approximately Month 10 (n=85,89,94) | -1.6 (14.46) | 0.0 (15.99) | 0.3 (12.61)
  Cycle 13 - approximately Month 13 (n=72,72,81) | -3.8 (15.61) | -1.0 (14.59) | 0.3 (12.60)
  Cycle 16 - approximately Month 16 (n=62,50,61) | -2.1 (14.95) | -2.9 (14.16) | -0.9 (12.23)

27. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13, 16 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) In Future Perspective Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. Questions used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale. For the future perspective scale, higher score = better perspective of the future.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=112,121,124) | 4.7 (23.74) | 4.3 (23.56) | 7.6 (22.38)
  Cycle 7 - approximately Month 7 (n=93,108,112) | 14.6 (24.45) | 7.7 (23.86) | 9.8 (20.62)
  Cycle 10 - approximately Month 10 (n=83,88,97) | 17.3 (27.84) | 6.6 (22.40) | 14.5 (21.73)
  Cycle 13 - approximately Month 13 (n=71,73,81) | 17.3 (27.15) | 6.3 (23.78) | 11.9 (24.67)
  Cycle 16 - approximately Month 16 (n=62,52,62) | 18.5 (25.30) | 7.7 (28.49) | 14.4 (26.62)

28. Secondary Outcome: Change From Baseline to Cycles 4, 7, 10, 13, 16 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) In Body Image Scale
Description: Data as of 11 May 2010 cutoff. EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. Questions used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale. For the body image scale, higher scores = better body image.
Time Frame: Baseline (Day 0), Months 4, 7, 10, 13, 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MPR+R | MPR+p | MPp+p
Number analyzed (Participants) | 152 | 153 | 154
units on a scale
  Cycle 4 - approximately Month 4 (n=110,117,119) | 2.1 (35.36) | -0.3 (37.27) | 4.5 (25.65)
  Cycle 7 - approximately Month 7 (n=88,104,108) | 3.8 (33.32) | 2.6 (37.94) | 5.2 (27.78)
  Cycle 10 - approximately Month 10 (n=79,83,94) | 7.6 (33.32) | -4.0 (43.69) | 3.9 (26.72)
  Cycle 13 - approximately Month 13 (n=68,72,79) | 1.0 (31.01) | -0.5 (44.23) | 5.1 (32.51)
  Cycle 16 - approximately Month 16 (n=59,52,61) | 3.4 (32.58) | 6.4 (41.25) | 2.7 (28.08)

ADVERSE EVENTS:
Time Frame: Up to 169 weeks (Double-blind therapy period plus 4 weeks)
Arm/Group | MPR+R | MPR+p | MPp+p
Serious Adverse Events (participants affected / at risk) | 66/150 | 62/152 | 56/153
Other Adverse Events (participants affected / at risk) | 149/150 | 151/152 | 152/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPR+R (N=150) | MPR+p (N=152) | MPp+p (N=153)
Pneumonia (Infections and infestations) | 4 (5) | 8 (9) | 8 (8)
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Norwalk virus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 8 (10) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 4 (5) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 2 (2) | 7 (8)
Fatigue (General disorders) | 4 (4) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3) | 5 (6)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (3) | 1 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 6 (7) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2)
Leukaemia plasmacytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Light chain disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2) | 4 (4)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (4) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Renal amyloidosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Oral intake reduced (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Monoclonal immunoglobulin present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPR+R (N=150) | MPR+p (N=152) | MPp+p (N=153)
Neutropenia (Blood and lymphatic system disorders) | 117 (951) | 116 (807) | 78 (398)
Anaemia (Blood and lymphatic system disorders) | 99 (417) | 91 (351) | 82 (293)
Thrombocytopenia (Blood and lymphatic system disorders) | 103 (514) | 100 (532) | 68 (268)
Leukopenia (Blood and lymphatic system disorders) | 54 (418) | 58 (449) | 49 (237)
Nausea (Gastrointestinal disorders) | 37 (65) | 39 (66) | 51 (93)
Constipation (Gastrointestinal disorders) | 49 (80) | 39 (66) | 37 (57)
Diarrhoea (Gastrointestinal disorders) | 43 (124) | 36 (62) | 37 (50)
Vomiting (Gastrointestinal disorders) | 15 (24) | 18 (27) | 19 (30)
Abdominal pain upper (Gastrointestinal disorders) | 13 (18) | 7 (9) | 13 (19)
Abdominal pain (Gastrointestinal disorders) | 16 (25) | 9 (9) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 12 (17) | 6 (6) | 8 (10)
Dry mouth (Gastrointestinal disorders) | 12 (14) | 7 (8) | 4 (6)
Fatigue (General disorders) | 46 (110) | 51 (97) | 57 (101)
Pyrexia (General disorders) | 32 (47) | 38 (63) | 27 (33)
Oedema peripheral (General disorders) | 30 (47) | 35 (59) | 25 (35)
Asthenia (General disorders) | 33 (67) | 22 (38) | 25 (39)
Oedema (General disorders) | 8 (11) | 14 (16) | 7 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 46 (96) | 45 (77) | 51 (76)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 17 (23) | 29 (38)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 (37) | 18 (22) | 21 (38)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (12) | 22 (28) | 17 (23)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 (34) | 17 (36) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (18) | 6 (11) | 10 (12)
Nasopharyngitis (Infections and infestations) | 23 (34) | 21 (32) | 26 (34)
Upper respiratory tract infection (Infections and infestations) | 16 (25) | 19 (23) | 15 (20)
Bronchitis (Infections and infestations) | 16 (25) | 15 (20) | 12 (16)
Urinary tract infection (Infections and infestations) | 12 (15) | 11 (15) | 11 (13)
Anorexia (Metabolism and nutrition disorders) | 24 (37) | 36 (54) | 23 (26)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (42) | 10 (32) | 17 (46)
Hypokalaemia (Metabolism and nutrition disorders) | 17 (21) | 12 (23) | 6 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 10 (12) | 8 (18) | 10 (25)
Dizziness (Nervous system disorders) | 15 (22) | 20 (21) | 16 (21)
Paraesthesia (Nervous system disorders) | 15 (19) | 10 (17) | 6 (7)
Headache (Nervous system disorders) | 11 (29) | 16 (26) | 21 (21)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (14) | 9 (13) | 5 (10)
Dysgeusia (Nervous system disorders) | 6 (9) | 10 (13) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 30 (62) | 42 (63) | 12 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (24) | 13 (16) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 34 (47) | 27 (33) | 21 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (34) | 15 (20) | 18 (22)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (15) | 7 (10) | 11 (16)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 9 (10) | 9 (11)
Blood creatinine increased (Investigations) | 12 (21) | 6 (13) | 17 (33)
Weight decreased (Investigations) | 8 (10) | 13 (18) | 9 (11)
Insomnia (Psychiatric disorders) | 17 (18) | 20 (23) | 22 (35)
Depression (Psychiatric disorders) | 9 (12) | 17 (18) | 10 (10)
Hypertension (Vascular disorders) | 4 (5) | 9 (11) | 13 (23)
Hypotension (Vascular disorders) | 10 (13) | 4 (4) | 10 (10)
Vertigo (Ear and labyrinth disorders) | 13 (23) | 10 (13) | 14 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon investigator submission of a publication or presentation to Celgene, Celgene shall complete its review within 60 days after receipt of the proposed publication or presentation. Upon Celgene's request, proposed publication or presentation will be delayed up to 90 additional days to enable Celgene to secure adequate intellectual property protection of property of Celgene that would be affected by such proposed publication or presentation.